CLINICAL TRIAL: NCT05349422
Title: Addressing Antihypertensive Medication Adherence Through EHR-enabled Teamlets in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-00133; R01HL156355 (NIH)
Record Dates: First submitted 2022-04-22; First posted 2022-04-27 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Blood Pressure; Medication Adherence
MeSH Terms: conditions — Medication Adherence | interventions — Electronic Health Records

STUDY DESIGN:
Intervention Model Description: The study trial will utilize a practice-level cluster-randomized design, with 1:1 randomization at 10 clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Electronic Health Record (EHR) Enabled Teamlets
- Usual Care Group (No Intervention): Usual Care Clinical Decision Support (CDS) Tools

INTERVENTIONS:
Behavioral: Electronic Health Record (EHR) Enabled Teamlets — The intervention consist of four components: 1) patients with hypertension will be automatically screened for low medication adherence using linked EHR-pharmacy data at the time of a PCP encounter; 2) MAs will deliver a validated, rapid, survey of common causes of non-adherence; 3) MAs and/or RNs will address barriers to adherence tailored to survey response, including delivery of brief health coaching based on motivational interviewing; and 4) PCPs will address specific barriers to adherence based on survey response.
  Arms: Intervention Group

SUMMARY:
The study team will conduct a cluster randomized control trial in 10 NYU primary care practices to assess the effectiveness and implementation of the multicomponent intervention on medication adherence and blood pressure control for patients who are non-adherent to antihypertensive medications.

ELIGIBILITY:
Inclusion Criteria:

Individuals:

1. Age>18 years
2. Presence of Hypertension as defined by either:

   1. Blood pressure ≥140/90
   2. Hypertension diagnosis
   3. Prescription for at least one antihypertensive medication
3. Outpatient clinic visit in the NYULH between 06/1/2022 and 12/31/2025

MAs, PCPs, LPNs, and RNs:

1. A clinician from an NYULH ambulatory practice location.

   a. Eligible clinicians include physicians, medical assistants, licensed practical nurses, and registered nurses.
2. Adult patients during appointments with eligible clinicians
3. Age > 18 years

Exclusion Criteria:

1. Patients who decline to be observed.
2. The study team has no specific exclusion criteria for patients in chart review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1726 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2025-05-11 (Actual)

PRIMARY OUTCOMES:
Average Number of Days Covered (PDC) as a Measure of Medication Adherence | Month 12
  The proportion of days covered (PDC) is used to estimate medication adherence by looking at the proportion of days in which a person has access to the medication, over a given period of interest

SECONDARY OUTCOMES:
Average Number of Days Covered (PDC) as a Measure of Medication Adherence | Month 18
  The proportion of days covered (PDC) is used to estimate medication adherence by looking at the proportion of days in which a person has access to the medication, over a given period of interest
Mean Systolic Blood Pressure | Month 12
Mean Systolic Blood Pressure | Month 18
Mean Diastolic Blood Pressure | Month 12
Mean Diastolic Blood Pressure | Month 18

CONTACTS AND LOCATIONS:
Overall Officials: Saul Blecker, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Saul.Blecker@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Blecker S, Schoenthaler A, Martinez TR, Belli HM, Zhao Y, Wong C, Fitchett C, Bearnot HR, Mann D. Leveraging Electronic Health Record Technology and Team Care to Address Medication Adherence: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2023 Jul 7;12:e47930. doi: 10.2196/47930. PMID 37418304
- [Background] Kharmats AY, Martinez TR, Belli H, Zhao Y, Mann DM, Schoenthaler AM, Voils CI, Blecker S. Self-reported adherence and reasons for nonadherence among patients with low proportion of days covered for antihypertension medications. J Manag Care Spec Pharm. 2023 May;29(5):557-563. doi: 10.18553/jmcp.2023.29.5.557. PMID 37121253
- [Derived] Martinez TR, Schoenthaler AM, Mann DM, Belli H, Bearnot HR, Lustbader I, Blecker S. Healthcare Professionals' Perspectives on Addressing Patients' Medication Adherence in Primary Care Settings. J Eval Clin Pract. 2025 Dec;31(8):e70322. doi: 10.1111/jep.70322. PMID 41308044
- [Derived] Blecker S, Mann DM, Martinez TR, Belli HM, Zhao Y, Ahmed A, Fitchett C, Wong C, Bearnot HR, Voils CI, Schoenthaler AM. Medication Adherence in Hypertension: A Cluster Randomized Clinical Trial. JAMA Cardiol. 2025 Sep 1;10(9):914-921. doi: 10.1001/jamacardio.2025.2155. PMID 40632527